CLINICAL TRIAL: NCT04792502
Title: BrUOG 401: A Phase 2 Study of Mosunetuzumab With Lenalidomide Augmentation as First-line Therapy for Follicular and Marginal Zone Lymphoma
Brief Title: Mosunetuzumab With Lenalidomide Augmentation as First-line Therapy for Follicular and Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 401
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-03

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Planned Therapy (Experimental)
  Interventions: Drug: Mosunetuzumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Mosunetuzumab — Administered subcutaneously by injection beginning with 5 mg and increasing to 45 mg.
Drug: Lenalidomide — Patients in the augmentation cohort will be dosed continuously, 10 mg orally once daily, with or without food.

SUMMARY:
BrUOG-401 is a prospective, single-arm, phase 2 trial of first-line therapy in adult patients with previously untreated FL or MZL. All patients will be assigned the same initial treatment plan, modified by interim response assessment (IRA) after Cycle 4. All patients will start treatment with four 21-day cycles (C1-4) of mosunetuzumab alone (using step-up dosing during C1), followed by IRA. Patients who achieve CR at IRA will continue with additional 4 cycles (C5-8) of mosunetuzumab. Patients who achieve PR at IRA will receive mosunetuzumab with lenalidomide augmentation during C5-8. Primary response assessment (PRA) will occur after C8. Patients who remain in PR at PRA will continue for additional 4 cycles (extended augmentation).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document and to comply with the study protocol procedures.
2. Age ≥18 years at the time of signing informed consent. Because no dosing or adverse event data are currently available on the use of mosunetuzumab in patients <18 years of age, they are excluded from this study.
3. Histologically confirmed diagnosis of:

   * follicular lymphoma (grade 1, 2, 3a, or not otherwise specified) or
   * marginal zone lymphoma (nodal, extranodal, or splenic), according to 2016 WHO classification and confirmed to express the CD20 antigen by immunohistochemistry or flow cytometry. Patients in whom definitive pathologic subtype of FL/MZL is undetermined due to limited biopsy material can be enrolled if in the investigator's opinion integrated clinicopathologic data are consistent with the eligible diagnosis.
4. Agreement to provide, if available, lymphoma tissue for correlative analyses.
5. At least one bi-dimensionally measurable nodal lesion, defined as >1.5 cm in its longest dimension, or one bi-dimensionally measurable extranodal lesion, defined as >1.0 cm in its longest diameter; with the exception of splenic MZL, which must be evaluable using the International SMZL Group criteria.
6. No prior systemic therapy for B-cell lymphoma, except for palliative corticosteroids; prior local therapy (surgery, radiation therapy, or antibiotics) is allowed.
7. Indication to start systemic therapy for lymphoma:

   * Patients with FL must meet one of the GELF criteria:

     * any mass ≥7 cm (except spleen);
     * at least 3 nodes >3 cm in diameter;
     * symptomatic spleen enlargement;
     * local symptoms or compromise of normal organ function due to tumor mass;
     * presence of ascites or pleural effusion;
     * presence of B symptoms (fever, night sweats, or unintentional weight loss of >10% over ≤6 months);
     * serum lactate dehydrogenase or beta-2-microglobulin above upper limit of normal;
     * cytopenias due to underlying lymphoma (i.e., absolute neutrophil count <1.0 × 109/L, hemoglobin <10 g/dL, and/or platelet count <100 × 109/L).
   * Patients with MZL must have an indication to start therapy as assessed by the investigator.
8. Performance status ECOG 0, 1, or 2.
9. Adequate hematologic function (unless due to underlying lymphoma as established by bone marrow involvement or splenomegaly):

   * hemoglobin ≥9 g/dL,
   * absolute neutrophil count ≥1.0 x 109/L,
   * platelet count ≥75 x 109/L.
10. Glomerular filtration rate (GFR) ≥40 mL/min/1.73m2 using the Mayo Quadratic Formula.
11. The effects of mosunetuzumab on the developing human fetus are unknown. For this reason and because lenalidomide used in this trial is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) and refrain from donating eggs or sperm throughout the treatment and for 3 months after the last dose of trial therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
12. Agreement to enroll in and comply with all local requirements of the REVLIMID® (lenalidomide) Risk Evaluation and Mitigation Strategy (REMS®) program for the purpose of lenalidomide acquisition.

Exclusion Criteria:

1. Grade 3b follicular lymphoma or transformed lymphoma.
2. Prior treatment with any anti-CD20 antibody or lenalidomide for lymphoma.
3. Prior stem cell transplantation (autologous or allogeneic) or prior solid organ transplantation.
4. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products.
5. Known NYHA class 3/4 congestive heart failure, LVEF <40%, myocardial infarction within 6 months prior to enrollment, unstable angina, or unstable arrhythmia.
6. Chronic obstructive pulmonary disease (COPD) requiring oral corticosteroids or chronic oxygen.
7. History of autoimmune disease, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, idiopathic pulmonary fibrosis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, granulomatosis with polyangiitis, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, with the exception of: hypothyroidism (on stable dose of thyroid replacement therapy), asthma managed with inhaled medications only; type 1 diabetes mellitus on stable insulin regimen, Sjögren syndrome, immune thrombocytopenia or autoimmune hemolytic anemia that does not require systemic therapy; dermatologic condition (including eczema, psoriasis, lichen simplex chronicus, or vitiligo) with skin manifestations with rash covering <10% of body surface area and not requiring treatment other than low-potency topical corticosteroids for >12 months prior to registration.
8. Use of any systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) with the exception of corticosteroid treatment using <10 mg/day prednisone or equivalent within 2 weeks prior to first treatment; a brief course of palliative corticosteroids at higher doses (prednisone up to 100 mg daily, for up to 7 days) is allowed, but must be completed at least 7 days before the first dose of mosunetuzumab.
9. Any of the following conditions:

   * active bacterial infection requiring antibiotics
   * known or suspected chronic active Epstein Barr virus (CAEBV) infection
   * history of hemophagocytic lymphohistiocytosis (HLH)
   * confirmed progressive multifocal leukoencephalopathy (PML)
   * known active EBV or CMV viremia
   * positive test for hepatitis B surface antigen (HBSAg). Patients with a positive total/IgG hepatitis B core antibody (HBcAb) may participate if hepatitis B virus (HBV) DNA is undetectable at screening, if they agree to take entecavir or tenofovir, and undergo periodic DNA testing
   * positive hepatitis C virus (HCV) antibody, unless a negative polymerase chain reaction (PCR) for HCV is documented
   * positive test for HIV.
10. Administration of a live, attenuated vaccine within 4 weeks before first mosunetuzumab dose or anticipation that such a live, attenuated vaccine will be required during the study.
11. Current or past history of CNS disease, including stroke, epilepsy, or CNS vasculitis, or an advanced neurodegenerative disease; with the exception of: stroke >2 years before registration without any residual neurologic deficits and no subsequent transient ischemic attacks; history of epilepsy with no seizures for >2 years and not using any antiepileptic therapy; well-controlled Parkinson's disease (with no need for a significant medication adjustment for > 6 months).
12. History of other malignancy that could affect compliance with the protocol or interpretation of results; patients with a curatively treated skin cancer, in situ cervical cancer, or another malignancy treated curatively with a documented remission >2 years before registration are eligible.
13. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks before the first dose of mosunetuzumab.
14. Clinically significant liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
15. Any major surgery within 4 weeks before the first dose of mosunetuzumab, other than lymph node biopsy for diagnosis.
16. Evidence of other significant or uncontrolled medical or psychiatric conditions that could affect compliance with the protocol.
17. Any of the following abnormal laboratory values within 14 days prior to first dose of mosunetuzumab:

    * AST or ALT >3x ULN
    * total bilirubin >2 x ULN (unless due to Gilbert syndrome with indirect hyperbilirubinemia only)
    * INR>1.5 x ULN without anticoagulation
    * PTT or APTT >1.5x ULN in the absence of lupus anticoagulant.
18. Any radiation therapy within 2 weeks prior to first dose of mosunetuzumab.
19. Pregnancy, breast-feeding, or prisoner status. Women of childbearing potential must have a negative pregnancy test within 2 weeks before first dose of mosunetuzumab, and must undergo repeat pregnancy testing during each cycle of lenalidomide therapy (see Inclusion Criterion 11).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | At the end of Cycle 8 (each cycle is 21 days)
  The rate of complete response at the time of primary response assessment (PRA).

SECONDARY OUTCOMES:
Progression Free Survival | Time of study registration through end of follow-up, approximately 5 years.
  PFS will be determined according to the guidance from the International Working Group. The following events will be counted for PFS: disease progression, disease recurrence, initiation of new line of therapy, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Olszewski, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Lifespan Cancer Insitute, Providence, Rhode Island